CLINICAL TRIAL: NCT00022711
Title: A Phase II Study of Temozolomide (SCH 52365) in the Treatment of Patients With Relapsed Small Cell Lung Cancer
Brief Title: Temozolomide in Treating Patients With Relapsed or Progressive Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FCCC-01020; NCI-G01-2005 (Other: NCI)
Record Dates: First submitted 2001-08-10; First posted 2003-01-27 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Lung Cancer
Keywords: recurrent small cell lung cancer; intermediate type small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Temozolomide (Experimental): Temozolomide 150mg/m2/day daily. Repeat cycles every 28days for maximum of six months
  Interventions: Drug: temozolomide

INTERVENTIONS:
Drug: temozolomide — 150 mg/m2/day Repeat cycles every 28 days following first daily dose of each cycle until toxicity or disease progression for a maximum of six months

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of temozolomide in treating patients who have relapsed or progressive small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of temozolomide, in terms of response rate and safety, in patients with relapsed or progressive small cell lung cancer.
* Determine the time to progression and overall survival in patients treated with this drug.
* Assess quality of life of patients treated with this drug.

OUTLINE: This is a multicenter study. Patients are stratified according to response to prior chemotherapy (chemosensitive at least 60 days after prior therapy vs chemoresistant less than 60 days after or progression during prior therapy).

Patients receive oral temozolomide once daily on days 1-7 and 15-21. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed prior to each course of chemotherapy, at 30 days after study completion, and then every 8 weeks thereafter.

Patients are followed at 30 days and then every 8 weeks thereafter.

PROJECTED ACCRUAL: A total of 37-79 patients (14-33 chemosensitive and 23-46 chemoresistant) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed relapsed or progressive small cell lung cancer

  * Classical or intermediate variant OR
  * Relapsed or progressive extrapulmonary small cell carcinoma of unknown origin
* Bidimensionally measurable disease

  * At least 1 cm by 1 cm by physical exam or radiologic exam
  * Outside prior radiation port unless clinical evidence of disease progression
* Previously radiated brain metastases allowed provided stable or improved

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* More than 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* SGOT/SGPT no greater than 3 times ULN (5 times ULN if liver metastases present)
* Alkaline phosphatase no greater than 5 times ULN

Renal:

* Creatinine no greater than 2 mg/dL

Other:

* HIV negative
* No AIDS-related illness
* No frequent vomiting or medical condition that would interfere with oral medication administration (e.g., partial bowel obstruction)
* No active nonmalignant systemic disease that would preclude study
* No other active invasive malignancy within the past year or concurrently requiring ongoing treatment
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception for at least 1 month before, during, and for at least 3 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior biologic therapy
* No concurrent immunotherapy
* No concurrent biologic therapy
* Concurrent epoetin alfa allowed

Chemotherapy:

* At least 4 weeks since prior chemotherapy
* No more than 1 prior continuous or discontinuous chemotherapy regimen for metastatic disease
* No other concurrent chemotherapy

Endocrine therapy:

* Concurrent hormonal therapy to boost appetite allowed (e.g., corticosteroids or medroxyprogesterone)

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy to 15% or more of bone marrow
* At least 1 week since prior radiotherapy to less than 15% of bone marrow
* No prior radiotherapy to 50% or more of bone marrow
* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* Recovered from prior therapy
* No other concurrent investigational drugs
* Concurrent pamidronate allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2002-01; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corey J. Langer, MD, Study Chair — Fox Chase Cancer Center
Locations (17):
- United States (17):
  - Hunterdon Regional Cancer Center, Flemington, New Jersey
  - Kimball Medical Center, Lakewood, New Jersey
  - South Jersey Regional Cancer Center, Millville, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital Burlington County, Mount Holly, New Jersey
  - Riverview Medical Center - Booker Cancer Center, Red Bank, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - St. Francis Medical Center, Trenton, New Jersey
  - Bon Secours-Holy Family Health System, Altoona, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Pinnacle Health Hospitals, Harrisburg, Pennsylvania
  - Conemaugh Memorial Hospital, Johnstown, Pennsylvania
  - Saint Mary Regional Center, Langhorne, Pennsylvania
  - Central Montgomery Medical Center, Lansdale, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Pottstown Memorial Regional Cancer Center, Pottstown, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania